CLINICAL TRIAL: NCT01454765
Title: Generation of Haploid Stem Cells From Human Germ Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: rmb-maza0001-ctil
Record Dates: First submitted 2011-10-16; First posted 2011-10-19 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Induced Pluripotent Stem Cells

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Germ cells and Stem cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sperm sample from healthy volunteers
  Interventions: Other: generation of stem cells

INTERVENTIONS:
Other: generation of stem cells — Collected germ cells will be cultured in medium. The germ cell cultures will be infected with reprograming factors. Rare colonies with characteristic stem cell morphologies will be expanded.
  Other Names: generation of stem cells from somatic haploid germ cells

SUMMARY:
Human cells are diploid (contain a double set of chromosomes). The diploid genome is complex and therefore limits genetic research approaches in biomedical models. To overcome this problem experimental generation of haploid stem cells has been done in animals. The investigators aim at generating haploid stem cells from human germ cells that are a useful tool in genetic research and screening.

DETAILED DESCRIPTION:
Human cells are diploid (contain a double set of chromosomes). The diploid genome is complex and therefore limits genetic research approaches in biomedical models. To overcome this problem experimental generation of haploid stem cells has been done in animal models. haploid cells are easier for genetic manipulations, such as knock-in and knock-out of genes, and therefore should make a better experimental model. The investigators aim at generating haploid stem cells from human haploid germ cells.

ELIGIBILITY:
Inclusion Criteria:

1. males over the age of 18 and under 50
2. no known chronic illness
3. not taking any chronic drugs

Exclusion Criteria:

1. females
2. males under 18 or over 50
3. any known chronic illness
4. taking chronic medications

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Patients donated samples | June 2011-November 2013
  No samples collected to date

SECONDARY OUTCOMES:
No secomdary outcome | June 2011 - November 2013

CONTACTS AND LOCATIONS:
Overall Officials: Itay Maza, M.D, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam medical center, Haifa
  - Weizmann institute of science, Rehovot